CLINICAL TRIAL: NCT03752255
Title: The Effects of Verbal and Visual Information Techniques on Anxiety in Impacted Third Molar Surgery
Brief Title: Verbal and Visual Information Techniques on Anxiety in Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Dilek Menziletoglu, Principle Investigator, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NEU2
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-11

CONDITIONS: Impacted Third Molar Tooth
Keywords: Video; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anxiety measurement method (Experimental): Before the operation, patients in the experimental group will fill the anxiety scales (DAS and STAI). Then patients will watch a video about impacted tooth. This video will include the complications that patients may face and what should be done after the procedure. After the watching the video, patients will fill the both DAS and STAI.
  Interventions: Other: Anxiety measurement method
- Control (Placebo Comparator): Before the operation, patients in the experimental group will fill the anxiety scales (DAS and STAI). The verbal information in detail will be given to the patients by the surgeon.This verbal information will include the complications that patients may face and what should be done after the procedure.
  Interventions: Other: Anxiety measurement method

INTERVENTIONS:
Other: Anxiety measurement method — Two different techniques (video or verbal information) will be examined about impacted third molar surgery.

SUMMARY:
The aim of this study was to evaluate preoperative anxiety levels using dental anxiety scale (DAS) and the Spielberger State-Trait Anxiety Inventory (STAI).

DETAILED DESCRIPTION:
This study will based on a prospective, observational investigation of two different patient education techniques about the effect of third molar removal on patients' anxiety level. A total of 240 patients will be divided into two groups.

Information about operation procedures and a recovery will be given verbally in group 1 and information about operation procedures and recovery will be given in group 2. Anxiety levels were assessed by using DAS and (STAI).Paired t-test or Wilcoxon test will be used for intra-group comparison of anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Impacted third molar (bone and mucosa retention, mesioangular position)
* Patients with any chronic disease and allergy

Exclusion Criteria:

* Pericoronitis
* Patients with visual impairment
* Patients with psychological disorders
* Smoking
* Pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
The anxiety levels will be examined using DAS and STAI. | first day
  first day

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menziletoglu, Dr, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Karatay, Turkey (Türkiye)